CLINICAL TRIAL: NCT04235933
Title: A Phase I, Open-label Study to Evaluate the Pharmacokinetics, and Pharmacodynamics of a Single Dose of Tai Ai Injection in Healthy Adult Chinese Subjects
Brief Title: A Phase I Study of TACI-antibody Fusion Protein Injection (RC18) in Healthy Adult Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18C015
Record Dates: First submitted 2020-01-06; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Healthy
MeSH Terms: interventions — RC-18

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tai Ai(RC18) 80mg (Experimental): ·Experimental: Tai Ai 80mg: Injection: subcutaneous injection on abdomen; Intervention:Biological: RC18
  Interventions: Biological: Tai Ai(RC18) 80mg
- Tai Ai(RC18) 160mg (Experimental): ·Experimental: RC18 160mg: Injection: subcutaneous injection on abdomen; Intervention:Biological: RC18
  Interventions: Biological: Tai Ai(RC18) 160mg
- RC18 240mg (Experimental): ·Experimental: RC18 240mg Injection: subcutaneous injection on abdomen; Intervention: Biological: RC18
  Interventions: Biological: RC18 240mg

INTERVENTIONS:
Biological: Tai Ai(RC18) 80mg — The patient received one treatment of RC18 80mg in the test group
  Arms: Tai Ai(RC18) 80mg
Biological: Tai Ai(RC18) 160mg — The patient received one treatment of RC18 160mg in the test group
  Arms: Tai Ai(RC18) 160mg
Biological: RC18 240mg — The patient received one treatment of RC18 240mg in the test group
  Arms: RC18 240mg

SUMMARY:
to evaluate the pharmacokinetics, and pharmacodynamics of a single dose of Tai Ai injection in healthy adult Chinese subjects

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent as applicable to participate in the study, age 18-55, inclusive, male: female=1:1;
2. Body mass index between 18.5-26 kg/m², inclusive, with a body weight ≥50 kg (male), ≥45 kg (female);
3. Considered "healthy" by the investigator. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, as well as a complete physical examination including vital signs, 12-lead ECG, X-ray examination, infectious disease examination, peripheral blood cell count, platelet aggregation and coagulation function, blood chemistry, urine routine and stool routine ( include occult blood);
4. An understanding, ability, and willingness to fully comply with study procedures and restrictions.

Exclusion Criteria:

1. History of any hematological, digestive system, respiratory, cardiovascular, renal, neurological, psychiatric disease, metabolic disorders or tumor, which could affect the action, absorption, or disposition of the investigational product, or clinical or laboratory assessments;
2. History of abnormal bleeding or coagulation disorders (e.g. easy bruising, gum bleeding, prolonged bleeding after tooth extraction, joint hemorrhage; anemia in recent 1 year caused by menorrhagia, postpartum hemorrhage, vitamin K deficiency, haemorrhagic diseases caused by acquired coagulation factor antibodies, trauma or post-operative bleeding, etc.);
3. Pregnant or lactating female during screening period; subjects and their partners did not agree to take effective contraceptive measures (such as intrauterine devices, contraceptives or condoms) throughout the study period and within 30 days after the end of the visit period;
4. History of allergic to therapeutic or diagnostic protein products, allergic to two or more drugs and/or non-drug factors; suffering from allergic diseases;
5. History of surgery within six months before signing the informed consent; Willing to undergo surgery within two weeks after the end of the trial (including cosmetic surgery, dental surgery, oral surgery, etc.);
6. Participated an investigational product in recent 3 months;
7. Current use of any prescription or over-the-counter (herbal, vitamins, or healthcare products). Current use is defined as use within 14 days or PK equivalent of 5 half-lives, whichever is longer;
8. History of Bleeding or donated more than 400ml blood 3 months before screening period, or plan to denote blood within 1 month after the trial;
9. Consume more tobacco or alcohol (≥14 units of alcohol per week: one standard unit contains 14g of alcohol, equals to 360ml of beer, 45ml of 40% liquor or 150ml of wine; smokers with more than 5 cigarettes per day.);
10. Consume excessive caffeine-containing beverages, foods that may affect drug metabolism within four weeks before signing informed consent: coffee (≥1100 mL per day), tea (≥2200 mL per day), cola (≥2200 mL per day), energy drinks (≥1100 mL per day), chocolate (≥510 g per day);
11. Positive HIV, HBsAg, Hepatitis C virus, Tubercle Bacillus antibody screen;
12. Researchers believe that there are other factors that are not suitable for participating in the experiment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
C-max | Day 0、Day 1、Day 2、Day 3、Day 5、Day 8、Day 15、Day 22、Day 29、Day 43、Day 57
  Maximum observed plasma concentration
T-max | Day 0、Day 1、Day 2、Day 3、Day 5、Day 8、Day 15、Day 22、Day 29、Day 43、Day 57
  Time to reach maximum observed plasma concentration
T1/2 | Day 0、Day 1、Day 2、Day 3、Day 5、Day 8、Day 15、Day 22、Day 29、Day 43、Day 57
  apparent terminal half-life
AUC0-t | Day 0、Day 1、Day 2、Day 3、Day 5、Day 8、Day 15、Day 22、Day 29、Day 43、Day 57
  area under the plasma concentration time curve from time 0 to the time of last observed quantifiable concentration
AUC0-∞ | Day 0、Day 1、Day 2、Day 3、Day 5、Day 8、Day 15、Day 22、Day 29、Day 43、Day 57
  Area under the plasma concentration-time curve from time 0 extrapolated to infinity

SECONDARY OUTCOMES:
Evaluation of AEs (adverse events).Through observing number of total AEs and number of subjects with AEs and other factors of AEs ，to evaluate the safety and tolerance of healthy subjects. | Day 0、Day 1、Day 2、Day 3、Day 5、Day 8、Day 15、Day 22、Day 29、Day 43、Day 57
  Occurrence of all adverse events from signing of informed consent through end of study treatment.
Evaluation of Vital Signs | Day 0、Day 1、Day 2、Day 3、Day 5、Day 8、Day 15、Day 22、Day 29、Day 43、Day 57
  Through observing the normal and abnormal conditions of axillary temperature to evaluate the safety and tolerance of healthy subjects. Axillary temperature's normal ：≥36 and ≤37°C. Clinical significance of abnormal values as judged by the investigator
Evaluation of Vital Signs | Day 0、Day 1、Day 2、Day 3、Day 5、Day 8、Day 15、Day 22、Day 29、Day 43、Day 57
  Through observing the normal and abnormal conditions of Pulse rate to evaluate the safety and tolerance of healthy subjects. Pulse rate's normal ：≥60 and ≤100. Clinical significance of abnormal values as judged by the investigator
Evaluation of Vital Signs | Day 0、Day 1、Day 2、Day 3、Day 5、Day 8、Day 15、Day 22、Day 29、Day 43、Day 57
  Through observing the normal and abnormal conditions of Blood pressure (both systolic and diastolic) to evaluate the safety and tolerance of healthy subjects. systolic pressure 's normal： ≥90 and ≤139 ； diastolic pressure's normal ：≥60 and ≤89. Clinical significance of abnormal values as judged by the investigator
Evaluation of Vital Signs | Day 0、Day 1、Day 2、Day 3、Day 5、Day 8、Day 15、Day 22、Day 29、Day 43、Day 57
  Through observing the normal and abnormal conditions of respiration to evaluate the safety and tolerance of healthy subjects. respiration's normal ：≥10 and ≤24. Clinical significance of abnormal values as judged by the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Zhijun Li, M.D., Principal Investigator — The First Affiliated Hospital of Bengbu Medical University; Huan Zhou, M.D., Principal Investigator — The First Affiliated Hospital of Bengbu Medical University
Locations (1):
- Remegen，ltd., Yantai, Shandong, China